CLINICAL TRIAL: NCT01764724
Title: Consumer Attitudes and Understanding of Low Sodium Claims on Food: An Analysis of Healthy and Hypertensive Individuals
Brief Title: Attitudes and Understanding of Sodium Claims on Food Labels
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Advance Foods and Materials Network (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Stroke Network (Other)
Responsible Party: Principal Investigator, Mary R. L'Abbé, Earle W. McHenry Professor, and Chair, Department of Nutritional Sciences, University of Toronto
Other Study IDs: 201103SOK-01
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: Attitudes and understanding of sodium claims; General canadian population
MeSH Terms: conditions — Hypertension; Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Canadian Consumer Monitor Panel: Canadian Consumer Monitor Panel is a online consumer monitor panel which answers surveys every 8-10 weeks about diet and health.
  Interventions: Behavioral: Mock package questionnaire

INTERVENTIONS:
Behavioral: Mock package questionnaire — Within a online questionnaire we exposed participants randomly to 4 mock packages differing only by the nutrition claim it carried and asked participants to answer several questions on attitudes and understanding after each mock package.

SUMMARY:
Sodium-related claims on food labels should help people find lower sodium food choices; however consumer attitudes and understanding of such claims are unknown.

The objective of this study was to evaluate: 1) the attitudes and understanding to different types of permitted sodium claims and 2) the effect of hypertension on responses to such claims.

ELIGIBILITY:
Inclusion Criteria:

* Primary grocery shoppers
* Canadian adults between the ages 20 to 69 years

Exclusion Criteria:

* Did not have an email address or have access to internet

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A subsection of the Canadian Consumer Monitor Panel - a national representative online consumer panel comprised of 30,000 Canadians
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response to survey questions measuring attitudes towards sodium claims using 5 point likert rating scales | On average the survey took 25 minutes to complete
  Within an online survey, participants were exposed to 4 mock soup packages that differed only by the claim it carried. After being exposed to each mock package, participants were asked to rate their perceived attractiveness, healthiness, credibility, usefulness of the tested sodium claims using 5 point likert scales. Participants were also asked to rate their purchasing intentions of the mock soup product with the different sodium claims.
Response to survey questions evaluating participants understanding of sodium claims | On average the survey took 25 minutes to complete
  After each mock package, understanding of sodium claims was evaluated using various survey methods. First, participants were asked to rate their perceived clarity of the wording of the claim using a 5 point likert scale (a subjective measure of understanding). Second, participants were ask to rate, on 5 point likert scales, the perceived benefit of consuming the mock package for subgroups with different health conditions (an indirect measure of understanding). Finally we asked participants, in an open ended question, to explain what a claim means to a friend (an objective measure of understanding).

CONTACTS AND LOCATIONS:
Overall Officials: Mary R L'Abbé, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Wong CL, Arcand J, Mendoza J, Henson SJ, Qi Y, Lou W, L'Abbe MR. Consumer attitudes and understanding of low-sodium claims on food: an analysis of healthy and hypertensive individuals. Am J Clin Nutr. 2013 Jun;97(6):1288-98. doi: 10.3945/ajcn.112.052910. Epub 2013 Apr 10. PMID 23576050